CLINICAL TRIAL: NCT03916432
Title: HELIOS China Registry: A Prospective, Single-arm, Multicenter Study to Evaluate the HELIOS Biodegradable Polymer Sirolimus-eluting Stent in a 'Real-World' Patient Population
Brief Title: HELIOS China Registry: Evaluation of the HELIOS Stent in a 'Real-World' Patient Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Beijing Luhe Hospital (Other); Cangzhou People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First Affiliated Hospital of Shantou University Medical College (Other); Western Central Hospital of Hainan Province (Unknown); Second Affiliated Hospital of Hainan Medical College (Unknown); Huizhou Municipal Central Hospital (Other); First People's Hospital of Yulin (Other); Shaanxi Armed Police Corps Hospital (Unknown); Xi'an No.3 Hospital (Other Government); Tang-Du Hospital (Other); Ankang Central Hospital (Other); General Hospital of Ningxia Medical University (Other); Cardiovascular Hospital of Ningxia Medical University (Unknown); First Affiliated Hospital of Xinjiang Medical University (Other); Kaifeng Central Hospital (Other); Xinyang Central Hospital (Other); People's Hospital of Zhengzhou University (Other); Zhoupu Hospital, Pudong New Area, Shanghai (Unknown); Shanghai Longhua Hospital (Unknown); Huangshan Shoukang Hospital (Unknown); First Affiliated Hospital of Southern Anhui Medical College (Unknown); First Affiliated Hospital of Harbin Medical University (Other); Harbin Medical University (Other); Third Affiliated Hospital of Qiqihar (Unknown); First Affiliated Hospital of Jiamusi University (Unknown); Harbin First Hospital (Unknown); The Second Hospital of Shenyang Medical College (Other); Yingkou Central Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ky20182050-1
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Interventional group (Experimental): HELIOS biodegradable polymer sirolimus-eluting stents
  Interventions: Device: HELIOS biodegradable polymer sirolimus-eluting stents

INTERVENTIONS:
Device: HELIOS biodegradable polymer sirolimus-eluting stents — HELIOS biodegradable polymer sirolimus-eluting stents

SUMMARY:
The study aims to evaluate the safety and efficacy of biodegradable polymer sirolimus-eluting coronary stent system (HELIOS) in patients with coronary artery disease . The primary endpoint is target lesion failure, a composite endpoint of cardiac death, target vessel related myocardial infarction and clinically-driven target lesion revascularization at 1 year follow-up.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm clinical registry investigating the safety and efficacy of biodegradable polymer sirolimus-eluting coronary stent system(HELIOS) in patients with coronary artery disease . The HELIOS (Kimley Medical, Shenzhen, China) completed biodegradable polymer sirolimus-eluting stent (SES) is a novel polylactic-co-glycolic acid (PLGA),polymer cobalt-chromium DES with titanium oxides (TiO) film as the tie-layer.In total, we plan to recruit 3000 patients (HELIOS)in real world setting. The patients will be followed clinically at 1-, 6- month and 1-, 3-, 5-year. All clinical data will be collected and managed by statistical center, clinical endpoint adjudication committee.

ELIGIBILITY:
Inclusion Criteria:

1）18-85 years old, male or non-pregnancy female; 2）Patients with coronary artery disease who match the indication of stent implantation; 3）Patients who can understand the nature of the study, agree to participate and accept clinical follow-up

Exclusion Criteria:

1. Patients who can not tolerate the material or medication in this study; Pregnancy or lactation women
2. Patients who had participated in another investigational drug or device trial that has not completed the primary endpoint;
3. Patients are, in the opinion of the investigator, unable to comply with the requirements of the study protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
target lesion failure (TLF) | 12 months
  a composite endpoint of cardiac death, target lesion related myocardial infarction, and/or target lesion revascularization

SECONDARY OUTCOMES:
Patient oriented composite endpoint | 1、6、12、36、60 months
  a composite endpoint of all cause death, all myocardial infarction and all revascularization
all cause death | 1、6、12、36、60 months
  including cardiac and non-cardiac death
cardiac death | 1、6、12、36、60 months
  death from cardiac cause
Myocardial infarction | 1、6、12、36、60 months
  All myocardial infarction (MI) data were reported based on extended historical definitions.MI was always considered a target vessel, unless there was documented proof that the infarction arose from the nontreated coronary artery.
Stent thrombosis | 1、6、12、36、60 months
  Stent thrombosis (ST) was defined according to Academic Research Consortium criteria
target lesion revascularization | 1、6、12、36、60 months
  TLR was defined as any repeat revascularization by PCI or CABG

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, MD, PhD, Study Director — First Affiliated Hospital，Fourth Military Medical University
Locations (1):
- Ling Tao, Xi’an, Shanxi, China

REFERENCES:
- [Result] Yuan F, Chen X, Song X, Wang D, Zhang Z, Li W, Li Z, Li H, Chen X, Huo Y, Wang L, Lu C, Lu Q, Xu B, Li W, Lyu S; HOPE Investigator. Novel completed biodegradable polymer sirolimus-eluting stent versus durable polymer sirolimus-eluting stent in de novo lesions: nine-month angiographic and three-year clinical outcomes of HOPE trial. Chin Med J (Engl). 2014;127(14):2561-6. PMID 25043067
- [Derived] He X, Liu Y, Yin Z, Li F, van Geuns RJ, Garg S, Onuma Y, Serruys PW, Gao C, Tao L. Mid-term outcomes of paclitaxel-coated balloon for de novo non-small coronary lesions: a pooled analysis. BMC Med. 2025 Oct 31;23(1):598. doi: 10.1186/s12916-025-04429-9. PMID 41174582
- [Derived] Zheng B, Liu Y, Zhang R, Yang W, Su F, Wang R, Chen D, Shen G, Qiu Y, Wang L, Chen C, Wu Z, Li F, Li J, Li C, Gao C, Tao L; HELIOS Investigators. A novel biodegradable polymer-coated sirolimus-eluting stent: 1-year results of the HELIOS registry. Chin Med J (Engl). 2023 Aug 5;136(15):1848-1854. doi: 10.1097/CM9.0000000000002324. PMID 37306407